CLINICAL TRIAL: NCT01994707
Title: Remote Ischemic Preconditioning of Human Myocardium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Principal Investigator, Marek Deja, MD PhD, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NCN-2012/07/B/NZ5/02549
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Coronary Artery Bypass Graft Triple Vessel; Apoptotic DNA Damage
Keywords: Remote ischemic preconditioning; Coronary artery bypass graft surgery; Troponin T; Apoptosis; Experimental; Cardioprotection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote ischemic preconditioning (Active Comparator): Left arm blood pressure cuff inflation for 5 min then deflation of cuff for 5 min- cycle repeated 3 times before coronary artery bypass grafting.
  Interventions: Procedure: Remote ischemic preconditioning
- Placebo (Placebo Comparator): Deflated cuff on arm for 30 minutes.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — Blood pressure cuff inflation
  Arms: Remote ischemic preconditioning
Procedure: Placebo — Deflated cuff on arm for 30 minutes.
  Arms: Placebo

SUMMARY:
The investigators aim to definitively show if human myocardium can be remotely preconditioned. In the writings there are no experiments that would prove that the remote preconditioning protocol effects on the higher protection of the human myocardial cells, against the ischemia-reperfusion injury.

120 patients referred for coronary artery bypass grafting (CABG) procedure with use of cardiopulmonary bypass are planned will be included to the research. Patients will be randomized (1:1) to one of two groups: remote preconditioning or "placebo" intervention. On the day of surgery, after induction of anesthesia remote preconditioning will be elicited by 3 cycles of 5min inflation (ischemia) and 5 min deflation (reperfusion) of blood pressure cuff on the right arm. In the control group the blood pressure cuff is going to be placed on the upper limb but the preconditioning protocol will not be carried out. On cannulation for CPB, right atrial appendage and myocardial biopsies of the left ventricular will be harvested. The investigators will study: (1) resistance of myocardium to hypoxia/reperfusion injury in in vitro experiments, assessed in isolated right atrial pectinate muscle trabeculae (2) induction of apoptosis and status of mitochondria in myocardium after the period of ischemia, and reperfusion in vitro (3) amount of myocardial necrosis in-vivo induced by period of ischemia and reperfusion during CABG as assessed by postoperative myocardial necrosis markers release (4) the systolic function of the myocardium at the postoperative and the kidney function in the postoperative period evaluated by the creatinine clearance; (5) induction of apoptosis and status of mitochondria in myocardium after the period of ischemia, and reperfusion during coronary artery bypass grafting, assessed in myocardial.

There is going to be an ability to define does the remote preconditioning influence on the occurrence of apoptosis in the human myocardium in the in vivo conditions and does it influence on the postoperative course in patients undergoing cardiac surgery procedures. The investigators will try to study if remote preconditioning modify induction of apoptosis and its structure in response to injury. In case the effect of remote preconditioning is not measurable in ex-vivo assessment, the future attempt at implementing this phenomenon in clinical practice may be futile and should not be continued until the effect can be confirmed in controlled experimental setting.

DETAILED DESCRIPTION:
The investigators will study:

1. Resistance of isolated right atrial pectinate muscle trabeculae to simulated hypoxia/reperfusion in functional organ bath model
2. Resistance of isolated right atrial pectinate muscle trabeculae to induction of apoptosis by simulated hypoxia/reperfusion
3. Resistance of mitochondria in isolated right atrial pectinate muscle trabeculae to changes induced by simulated hypoxia/reperfusion

Simultaneously we will assess:

1. Amount of myocardial necrosis in vivo induced by period of ischemia and reperfusion during coronary artery bypass grafting (CABG) as assessed by postoperative myocardial necrosis markers release profile
2. Myocardial function in vivo after the period of ischemia and reperfusion during CABG as assessed by hemodynamic measurements (thermodilution method), oxygen supply/consumption and inotropic support requirements
3. Induction of apoptosis and status of mitochondria after the period of ischemia, and reperfusion during CABG as assessed in left ventricular myocardial biopsies The investigators will try correlate the in vitro and in vivo findings from the same patients.

Methodology The study will be conducted both in vivo and ex-vivo. Patients referred for CABG for stable coronary artery disease will be recruited and randomized (1:1) by random digit generator to one of two groups: remote preconditioning or "placebo" intervention. Only patients in who at least 3 coronary artery bypass grafts with use of cardiopulmonary bypass (CPB) are planned will be included. On the day of surgery, after induction of anesthesia and before the skin incision remote preconditioning will be elicited. The "placebo" group will have the pressure cuff placed on the right arm but no inflations will be performed. To obtain blinding, the inflations will occur under surgical drapes, and will be performed by the same person every time, who will be involved in random sequence generation, and remote preconditioning application, but not in the care of the patient, or other research related tasks.

All consented patients will have preoperative echocardiography, electrocardiography and blood tests including fool blood count, creatinine, BUN, and liver function test performed as part of their routine preoperative care. Additionally troponin T and CK-MB levels will be assessed. Furthermore patients will have performed electrocardiography on 1st day after operation.

Anesthesia will be standardized and consist of midazolam 15mg orally 1h before surgery, etomidate 0.2mg/kg, fentanyl 5g/kg and pancuronium 0.1mg/kg iv for anesthesia induction, propofol 0.5-1.0 mg/kg/h and fentanyl 4g/kg/h infusion for anesthesia maintenance. No anesthetic gases will be used. Full hemodynamic monitoring will be used with Swan-Ganz catheter (not routine in CABG patients). First hemodynamic measurements and oxygen supply/consumption calculations will be performed preoperatively.

Functional in vitro assessment. On cannulation for CPB, right atrial appendage, which is routinely removed and discarded for venous cannula placement will be harvested in all patients. The tissue will be was transferred in ice cold Krebs-Henseleit solution to the isolated organ laboratory in our department. One pectinate muscle trabecula will be harvested for baseline assessment of apoptosis or mitochondria (see below). Another single trabecula less than 1mm in diameter will be mounted in the organ chamber - Schuler Organbath (Hugo Sachs Elektronik, March-Hugstetten, Germany (HSE)) containing Krebs-Henseleit solution. It will be oxygenated via glass frit with carbogen (95% oxygen, 5% carbon dioxide) and maintained at 37°C. The trabecula will be driven with 1Hz 50ms square stimuli using platinum field electrodes and the potential of 150% of the threshold for given preparation. The stimulator Type 215 (HSE) will be used. The contraction force will be measured with F30 isometric force transducer Type 372 (HSE). The signal will be enhanced with TAM A PlagSYS transducer amplifier module Type705 (HSE) and recorded using PowerLab/4SP system and Chart software (AD Instruments).

The trabecula will be gradually stretched to 90% of optimal tension according to Frank-Starling relationship and left for 30min of stabilization and washout.

60min ischemia will be simulated by substituting oxygen in carbogen with argon (95% argon, 5% carbon dioxide) and replacing Krebs-Henseleit solution with one containing no glucose or pyruvate. On reoxygenation the carbogen will be added again and the tissue bath solution will be replaced with one used initially. The tissue will be was washed several times and left for 120min of reoxygenation period with washout every 15 min. This functional model of hypoxia reoxygenation has been used in our laboratory before [12-14]. Replacement of oxygen with argon results in the drop of tissue bath oxygen partial pressure from 475±52mmHg to 51±1.8mmHg (p<0.001) [37-39]. It is accompanied by significant and rapid decline in isometric contraction force. During reoxygenation the contraction force returns initially and next we observe slow decline of muscle inotropism which we interpret as development of reoxygenation injury. At the end, we will use 10-4 M norepinephrine ((-)-Arterenol Bitartrate) to test for stunning.

The contraction force will be recorded continuously. Contractility will be expressed in percent of the initial contraction force for given preparation. The investigators will compare the maximal recovered contraction force, the contraction force after 30min and 120min of reoxygenation and the contraction force produced by adding 10-4M norepinephrine at the end of reoxygenation.

The investigators will also look for the signs of ischemic contracture development defined as an increase of resting tension of the trabecula. This increase, if present, starts shortly after the onset of hypoxia and continues steadily throughout the whole hypoxia period. The investigators will compare the increase in resting tension (in mN/mg tissue mass) at the end of hypoxia, that is at the time of maximal contracture.

All measurements, and in particular recovery of function will be compared between trabeculae from remotely preconditioned and "placebo" patients.

Two atrial trabeculae from the same appendage, one harvested at baseline, and another subjected to functional experiment (60 min hypoxia + 120 min reoxygenation) will be studied each time for:

* apoptosis induction - Caspase 3 and cleaved Caspase 3, PARP and cleaved PARP expression measured with Western-Blot, or
* apoptosis induction - assessed with TUNEL and immunohistochemistry staining for Caspase 3, cleaved Caspase 3, PARP and cleaved PARP, or
* state of mitochondria (electron microscopy) As we plan to randomize 120 patients (see below) the material for apoptosis and mitochondria studies will be randomly taken from 60 patients (30:30) for Western Blot, 40 patients (20:20) for immunohistochemistry and TUNEL, and 20 patients (10:10) for electron microscopy.

Western Blot (2 trabeculae, baseline and after hypoxia/reoxygenation, from 30 remotely preconditioned and 30 "placebo" patients).

For Western Blot immunoassay the trabeculae will be placed in liquid nitrogen Immunohistochemistry (2 trabeculae, baseline and after hypoxia/reoxygenation, from 20 remotely preconditioned and 20 "placebo" patients).

Expression of Caspase 3, cleaved Caspase 3, PARP and cleaved PARP proteins in tissue sections will be detected immunohistochemically. Trabeculae will be fixed overnight in 10% neutral-buffered formalin (phosphate buffer), subsequently passed through graded alcohol solutions, processed three times in xylene, and finally embedded in paraffin blocks. The documentation of immunohistochemical reactions will be performed with SSC-DC58AP camera (Sony) coupled with Nikon Eclipse E400 optical microscope.

TUNEL (terminal deoxynucleotidyl transferase dUTP nick and labeling) (2 trabeculae, baseline and after hypoxia/reoxygenation, from 20 remotely preconditioned and 20 "placebo" patients).

Tissue sections will be deparaffinized in 2 changes of xylene for 5 minutes each, and hydrated with 2 changes of 100% ethanol for 3 minutes each, and 95% ethanol for 1 minute. The documentation of immunohistochemical reactions will be performed with SSC-DC58AP camera (Sony) coupled with Nikon Eclipse E400 optical microscope.

Electron microscopy (2 trabeculae, baseline and after hypoxia/reoxygenation, from 10 remotely preconditioned and 10 "placebo" patients).

Trabeculae will be placed in cacodyl buffer with 2% glutaraldehyde. The mitochondria will be micrographed with JEOL-JEM 100CX transmission electron microscope (JEOL Inc, Peabody, Mass) with magnification x16000. The electron micrographs will next be saved and mitochondria size and structure will be analyzed using Image ProPlus software (Media Scanalytics).

The in vivo trial The operation will be performed with the use of CPB in normothermia by experienced cardiac surgeon. Intermittent warm-blood (37°C) antegrade cardioplegia (miniplegia) will be used for myocardial protection. As only patients requiring at least 3 coronary bypass grafts will be recruited, we expect aortic crossclamp time to last at least 30 minutes. After cross clamp removal the proximal anastomoses will be performed using side biting clamp. The patient will be weaned off CPB, hemostasis will be secured and the chest will be closed over chest tubes. Just before closing the chest 16G needle-true cut biopsy of the left ventricular myocardium will be obtained from the apex area. The investigators expect the reperfusion time from the cross-clamp removal to obtaining the biopsy to last at least 40 min. The exact ischemia (cross-clamp) time, and reperfusion time (until obtaining the biopsy) will be measured.

The myocardial biopsies will be harvested and assessed in the same way as atrial trabecule. The investigators will randomly perform Western blotting in 60 (30:30) biopsies harvested on liquid nitrogen, immunohistochemistry including TUNEL in 40 (20:20) harvested on 10% neutral buffered formalin, and electron microscopy in 20 (10:10) harvested on cacodyl buffer with 2% glutaraldehyde. The methods of assessing Caspase3, cleaved Caspase 3, PARP, cleaved PARP, TUNEL and mitochondria have been described above.

After the operation patient will be transferred to ICU and treated as per routine.

The primary endpoint of clinical observation will be the postoperative release of cardiac troponin T.

The investigators will measure serum concentration of cardiac Troponin T (electrochemiluminescence "ECLIA", Roche) preoperatively and next 72h from cross-clamp removal. At the same time points the level of creatine kinase isoenzyme MB will be assessed (enzymatic assay, Roche). The area under the curve of the marker level over time will be compared between the groups.

To assess the myocardial function all patients will have pulmonary artery catheter (Swan Ganz catheter) inserted preoperatively. Full hemodynamic assessment (thermodilution method) as well as oxygen metabolism status based on arterial and mixed venous gas analysis will be performed preoperatively and next 48h after aortic cross-clamp removal.

Apart from measuring cardiac index we will calculate left and right cardiac work indices. The oxygen delivery index and extraction ratio will be calculated. The lactate levels will also be measured. The investigators will also assess the need for inotropic support at the same time points using so called inotropic index.

All patients will have postoperative electrocardiogram on day 2 and 4 as per postoperative care routine and additionally on 1st day after operation. Similarly other routine postoperative tests that are performed as part of the routine postoperative care will be performed, monitored and used to look for the differences in postoperative course. This includes echocardiography as well as creatinine (eGFR).

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders.
2. Patients with stable coronary artery disease referred for surgical revascularization in who at least 3 coronary artery bypass grafts are planned with use of cardiopulmonary bypass.

Exclusion Criteria:

1. Age below 18 and above 80.
2. Plan to use radial artery as a graft.
3. Plan to perform other concomitant cardiac procedure in addition to CABG.
4. Diabetes mellitus.
5. Troponin T level before surgery in excess of 99th percentile of upper reference limit.
6. Acute coronary syndrome in last 14 days before surgery.
7. Angina pectoris in last 48 hours before surgery.
8. Significant peripheral vascular disease.
9. Renal disease with either creatinine level ≥ 2mg/dl or estimated glomerular filtration rate < 30ml/h/1.73m2.
10. Renal replacement therapy.
11. Clinically relevant hepatic insufficiency with bilirubin level at least 1.5 times above upper limit of normal or AlAT, AST levels at least 2 times above upper limit of normal.
12. Advanced lung disease with FEV1 < 40% of predicted value.
13. Severe systolic dysfunction of left ventricle (EF<35%).
14. Pregnancy.
15. Psychiatric disease.
16. Drug or alcohol abuse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2013-08; Primary Completion 2016-01-10 (Actual); Study Completion 2016-04-27 (Actual)

PRIMARY OUTCOMES:
Troponin-T | 72 hours
  Troponin-T release over the perioperative 72-hour period and its area under the curve (AUC)

SECONDARY OUTCOMES:
Creatine Kinase isoenzyme MB, full hemodynamic assessment with oxygen metabolic assessment and creatinine clearance (CKD-Epi method) | 1 week post surgery
Resistance of isolated right atrial pectinate muscle trabeculae to simulated hypoxia/reperfusion in functional organ bath model. | Day 1 of the RICP intervention
  All measurements, and in particular recovery of function will be compared between trabeculae from remotely preconditioned and "placebo" patients.
Resistance of isolated right atrial pectinate muscle trabeculae to induction of apoptosis by simulated hypoxia/reperfusion. | 1day at the moment of harvesting
  Two atrial trabeculae from the same appendage, one harvested at baseline, and another subjected to functional experiment (60 min hypoxia + 120 min reoxygenation) studied for:
  * apoptosis induction (Caspase 3 and cleaved Caspase 3, PARP and cleaved PARP -Western-Blot) or
  * apoptosis induction (Caspase 3, cleaved Caspase 3, PARP, cleaved PARP immunohistochemistry, TUNEL) or
  * state of mitochondria (electron microscopy)
Induction of apoptosis and status of mitochondria after the period of ischemia, and reperfusion during coronary artery bypass grafting as assessed in left ventricular myocardial biopsies. | 1 day at the moment of harvesting
  LV myocardium studied for:
  * apoptosis induction (Caspase 3 and cleaved Caspase 3, PARP and cleaved PARP -Western-Blot) or
  * apoptosis induction (Caspase 3, cleaved Caspase 3, PARP, cleaved PARP immunohistochemistry, TUNEL) or
  * state of mitochondria (electron microscopy)
Alveolar-arterial gradient (A-a gradient), S100 concentration, NGAL and zonulin concentration | 1st week post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marek A. Deja, MD PhD, Principal Investigator — Medical University of Silesia
Locations (1):
- Medical University of Silesia, Katowice, Poland

REFERENCES:
- [Derived] Deja MA, Piekarska M, Malinowski M, Wiaderkiewicz R, Czekaj P, Machej L, Weglarzy A, Kowalowka A, Kolodziej T, Czech E, Plewka D, Mizia M, Latusek T, Szurlej B. Can human myocardium be remotely preconditioned? The results of a randomized controlled trial. Eur J Cardiothorac Surg. 2019 Jun 1;55(6):1086-1094. doi: 10.1093/ejcts/ezy441. PMID 30649238
- [Derived] Deja MA, Wiaderkiewicz R, Czekaj P, Czech E, Malinowski M, Machej L, Weglarzy A, Kowalowka A, Piekarska M, Szurlej B, Latusek T. Remote Ischaemic PrEconditioning of Human Myocardium (RIPE): study protocol for a double-blinded randomised controlled trial. Kardiol Pol. 2018;76(1):136-143. doi: 10.5603/KP.a2017.0180. Epub 2017 Oct 5. PMID 28980297